CLINICAL TRIAL: NCT01527279
Title: Clinical Efficacy of Antazoline in Rapid Cardioversion of Paroxysmal Atrial Fibrillation - a Single Centre, Randomized, Double-blind, Placebo-controlled Study (the AnPAF Study)
Brief Title: Antazoline in Rapid Cardioversion of Paroxysmal Atrial Fibrillation
Acronym: AnPAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Antazoline
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: atrial fibrillation; paroxysmal; cardioversion; antazoline
MeSH Terms: conditions — Atrial Fibrillation | interventions — Antazoline; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Any patient fulfilling the inclusion criteria will be prepared to pharmacological cardioversion in a standard way comprising of standard baseline 12-lead ECG, continuous ECG monitoring, periodic noninvasive blood pressure monitoring (BP) and iv line. After drug administration the patient will be observed for 1.5 hour after the last dose with exit ECG and BP measure taken at the end of observation. Further treatment of the patient depends on clinical state and follows appropriate clinical guidelines.
  Interventions: Drug: 0.9% saline
- Antazoline (Experimental): Any patient fulfilling the inclusion criteria will be prepared to pharmacological cardioversion in a standard way comprising of standard baseline 12-lead ECG, continuous ECG monitoring, periodic noninvasive blood pressure monitoring (BP) and iv line. After drug administration the patient will be observed for 1.5 hour after the last dose with exit ECG and BP measure taken at the end of observation. Further treatment of the patient depends on clinical state and follows appropriate clinical guidelines.
  Interventions: Drug: antazoline

INTERVENTIONS:
Drug: antazoline — Patients assigned to antazoline group will be administered antazoline in boluses of 50mg diluted to 10cm3 every 5 minutes up to cumulative dose of 250mg or conversion of AF to SN. Drug administration will also be stopped in case of serious adverse event or conversion of AF to different supraventricular arrhythmia. BP will be measured before every injection.
  Other Names: Phenazolinum
  Arms: Antazoline
Drug: 0.9% saline — Patients assigned to control group will be administered 0.9% saline in boluses of 10cm3 every 5 minutes up to cumulative volume of 50cm3, conversion of AF to SN or in case of serious adverse event or conversion of AF to different supraventricular arrhythmia. BP will be measured before every injection.
  Arms: Placebo

SUMMARY:
The purpose of this randomized, double blind, placebo-controlled, superiority clinical trial was to assess clinical efficacy of antazoline in rapid conversion of atrial fibrillation during observation sinus rhythm.

DETAILED DESCRIPTION:
Antazoline is a first generation antihistaminic agent with chinidin-like properties. When administered intravenously, antazoline exerts a strong antiarrhythmic effect on supraventricular arrhythmia especially on atrial fibrillation (AF) facilitating rapid conversion to sinus rhythm. Despite relative lack of published data antazoline is marketed in Poland and widely used in cardiology wards and emergency rooms due to its efficacy, safety and rapid onset of action within minutes of administration.

To show superiority of antazoline over placebo a sample size of 80 patients was calculated based on following assumptions: two-tailed test, a type I error of 0.01, a power of 90%, efficacy of placebo 5%, efficacy of antazoline 50% and 20% drop-out rate to fulfill the criteria of intention-to-treat analysis. Due to presumed lack of statistical power the secondary end points and safety endpoints will be considered exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for participating in the study and written standard version of informed consent for cardioversion accepted in Institute of Cardiology, Warsaw, Poland
* Age above 18 and good general condition
* Potassium level over 3.5 mmol/l
* Stable cardio-pulmonary state on enrollment
* In case of unclear history of heart failure or suspicion of impaired left ventricle function echocardiography is indicated prior to enrollment
* A long-term antiarrhythmic drug therapy is allowed

Exclusion Criteria:

* Lack of written informed consent
* Antazoline allergy
* AF related to significant valvular disease
* Clinically significant heart failure or ejection fraction < 55%
* Diastolic blood pressure (BP) < 100mmHg
* History of significant bradyarrhythmia not treated with permanent pacemaker
* QT prolongation over 440ms or QTc (Bazett's formula) over population norm
* Tachycardia > 160'
* Advanced liver or kidney failure
* Acute coronary syndrome, coronary artery by-pass graft, stroke or transient ischemic attack within 30 days before enrollment
* Preexcitation in ECG not treated by radiofrequency ablation of accessory pathway
* Signs and symptoms of ischemia related to AF
* An investigational drug used within 30 days before enrollment
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-11; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Conversion of AF to SN confirmed in standard 12-lead ECG during observation period after first iv bolus | 1.5 hour

SECONDARY OUTCOMES:
Time to conversion of AF to SN | 1.5 hour
  in minutes since first injection
Return of AF during observation period | 1.5 hour
Serious adverse event defined as every adverse event requiring hospitalization or prolonged observation | 1.5 hour
Arterial pressure < 90mmHg | 1.5 hour
Disturbances of atrio-ventricular conduction | 1.5 hour
Sustained supraventricular arrhythmia other than AF | 1.5 hour
New complex ventricular arrhythmia | 1.5 hour
  Ventricular arrhythmia other than premature ventricular contraction
Hot flush | 1.5 hour
Drowsiness | 1.5 hour
Headache | 1.5 hour
Nausea/ vomiting | 1.5 hour
Chest pain | 1.5 hours
Tachycardia >180' | 1.5 hours
Prolongation of QTc in ms (Bazett's formula) in comparison to baseline | 1.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Szwed, MD, PhD, Study Chair — National Institute of Cardiology, Warsaw, Poland; Aleksander Maciag, MD, PhD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Michal M Farkowski, MD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, II Dept. of Coronary Heart Disease, Warsaw, Poland

REFERENCES:
- [Background] Farkowski MM, Maciag A, Dabrowski R, Pytkowski M, Kowalik I, Szwed H. Clinical efficacy of antazoline in rapid cardioversion of paroxysmal atrial fibrillation--a protocol of a single center, randomized, double-blind, placebo-controlled study (the AnPAF Study). Trials. 2012 Sep 11;13:162. doi: 10.1186/1745-6215-13-162. PMID 22967497
- [Derived] Maciag A, Farkowski MM, Chwyczko T, Beckowski M, Syska P, Kowalik I, Pytkowski M, Wozniak J, Dabrowski R, Szwed H. Efficacy and safety of antazoline in the rapid cardioversion of paroxysmal atrial fibrillation (the AnPAF Study). Europace. 2017 Oct 1;19(10):1637-1642. doi: 10.1093/europace/euw384. PMID 28339554